CLINICAL TRIAL: NCT05590520
Title: A Comparison of Injections of Botulinum Toxin and Topical Nitroglycerin Ointment for the Treatment of Chronic Anal Fissure :A Randomized Controlled Trial
Brief Title: Comparison of Injections of Botulinum Toxin and Topical Nitroglycerin Ointment for the Treatment of Chronic Anal Fissure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, Mubashra Badar, Resident, Pak Emirates Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIS 1cpsp
Record Dates: First submitted 2022-10-14; First posted 2022-10-21 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Fissure in Ano
Keywords: Fissure, botulinum toxin, Gtn ointment
MeSH Terms: conditions — Fissure in Ano

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum group (Experimental): The internal anal sphincter to be palpated and injected with a 27-gauge needle while the patient lying on his or her left side. Each patient will receive 0.4 ml of solution containing botulinum toxin (for a total of 20 U), administered as two injections of equal volume (0.2 ml), one on each side of the anterior midline of the internal anal sphincter. No sedation or local anesthesia to be used during the procedure)
  Interventions: Procedure: Botulinum injection
- GTN group (Active Comparator): 0.2 percent nitroglycerin ointment applied twice daily for six weeks.
  Interventions: Drug: GTN OINTMENT

INTERVENTIONS:
Procedure: Botulinum injection — Botox injection to be injected in internal anal sphincter to see the curative response in comparison to gtn cream application
  Other Names: Botox inj
  Arms: Botulinum group
Drug: GTN OINTMENT — 0.2%GTN applied on anal canal.
  Other Names: 0. 2% GTN
  Arms: GTN group

SUMMARY:
Patients will be randomized to receive treatment with either a total of 20 U of botulinum toxin(diluted in saline to a concentration of 50 U per milliliter.

DETAILED DESCRIPTION:
Lateral internal sphincterotomy, the most common treatment for chronic anal fissure, may cause permanent injury to the anal sphincter, which can lead to fecal incontinence. We compared two nonsurgical treatments that avert the risk of fecal incontinence.treatment with either topical nitroglycerin or botulinum toxin is effective as an alternative to surgery

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis: evidence of posterior circumscribed ulcer, with a large sentinel tag of skin, induration at the edges, and exposure of the horizontal fibers of the internal anal sphincter
* symptoms (post-defecatory or nocturnal pain, bleeding, or both) lasting for more than two months.

Exclusion Criteria:

* Patients with acute fissure
* fissure associated with other conditions (i.e., inflammatory bowel diseases, HIV infection, hemorrhoids, fistula in ano, anal abscesses, or anal or perianal cancer)
* those who had undergone previous surgical procedures in the anal canal.
* known hypersensitivity to component of the formulations of type A BTX
* pregnant or breast-feeding women 6-refusal of consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Healing of fissure | Within 6 weeks
  All the patients will undergo a pretreatment evaluation that will include clinical inspection of the fissure based on evidence of posterior circumscribed ulcer, with a large sentinel tag of skin, induration at the edges, and exposure of the horizontal fibers of the internal anal sphincter and symptoms including post-defecatory or nocturnal pain, bleeding, or both. Then they will be randomized to receive treatment with either botulinum toxin or 0.2 percent nitroglycerin ointment applied twice daily for six weeks. The outcome in each group will be evaluated clinically.The end point of the study would be complete healing after treatment. The treatment will be considered successful if the fissure healed. Persistence of the fissure in the absence of symptoms will be considered as symptomatic improvement.The Secondary endpoints will measurement of post defecatory pain on Visual analogue scale (VAS) at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mubashra Badar, Principal Investigator — Resident
Locations (1):
- Pak-Emirates Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
I'll publish the article and all data will be available for researchers
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available once published and will also be available as open source review
Access Criteria: All researchers will be allowed to buildup on this research.